CLINICAL TRIAL: NCT06334692
Title: Autoantibodies Against-nephrin in Idiopathic Nephrotic Syndrome
Acronym: BLINDER
Status: Recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: BLINDER
Record Dates: First submitted 2024-03-15; First posted 2024-03-28 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-05

CONDITIONS: Nephrotic Syndrome
Keywords: Idiopathic nephrotic syndrome; Minimal change disease; Focal segmental glomerulosclerosis; Permeability factor(s); B cells; Nephrin autoantibodies
MeSH Terms: conditions — Nephrotic Syndrome; Nephrosis, Lipoid; Glomerulosclerosis, Focal Segmental

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Sera from patients with biopsy-proven idiopathic MCD or FSGS who provided consent to store their samples in the certified biobank (Mario Negri Biological Resources Centre - Rare Diseases and Renal Diseases Biobank - CRB). Serum samples will be tested for the levels of anti-nephrin autoantibodies by in-house ELISA and results confirmed by commercial ELISA kits.
  Interventions: Diagnostic Test: In-house ELISA, and ELISA kits from "DBA Italy" (Abbexa).
- Controls: Sera from patients with biopsy-proven idiopathic membranous nephropathy who provided consent to store their samples in the certified biobank (Mario Negri Biological Resources Centre - Rare Diseases and Renal Diseases Biobank - CRB). Samples will be tested for the levels of anti-nephrin autoantibodies by in-house ELISA and results confirmed by commercial ELISA kits.
  Interventions: Diagnostic Test: In-house ELISA, and ELISA kits from "DBA Italy" (Abbexa).

INTERVENTIONS:
Diagnostic Test: In-house ELISA, and ELISA kits from "DBA Italy" (Abbexa). — "Nunc MaxiSorp" ELISA plates will be coated with recombinant extracellular domain of human nephrin. Patient serum samples will be added in appropriate dilution. Plates will be then incubated with biotin-conjugated anti human IgG antibody followed by incubation with horseradish peroxidase (HRP)-avidin conjugate. Then tetramethylbenzidine substrate will be added, and absorbance read at 450 nm.

SUMMARY:
This retrospective study is aimed at evaluating the levels of circulating anti-nephrin autoantibodies in patients with INS, including those with MCD/FSGS and in patients who have experienced relapse of FSGS post-transplant, compared to those of a control group of patients with nephrotic syndrome due to primary membranous nephropathy (MN).

DETAILED DESCRIPTION:
Nephrotic syndrome (NS) is one of the major "unsolved problems" in nephrology and represents a long-standing challenge in terms of pathogenetic mechanisms and the search for an effective cure.

Nephrotic-range proteinuria (>3.5 g/day) is accompanied by a set of abnormalities collectively known as NS. It is characterized by systemic complications resulting from alterations in the composition of the body's protein pool, sodium retention, dyslipidemia, coagulation factor abnormalities and a variable degree of renal failure. When secondary causes cannot be identified, the clinical presentation is called idiopathic nephrotic syndrome (INS). INS is associated with disappearance of podocyte pedicels (visible under the electron microscope) and minimal changes (minimal change disease, MCD) or, at the more advanced stage, focal segmental glomerulosclerosis (FSGS) under the light microscope. INS can be treated with corticosteroids, which represent the first-line treatment, however, among the forms of NS, FSGS has the lowest rate of response to therapy. More importantly, in 30% of patients with FSGS, disease recurrence develops rapidly after transplantation, sometimes within minutes or hours, and leads to the immediate onset of proteinuria and graft dysfunction. For post-transplant FSGS recurrence, no prevention or treatment strategies are available and current therapeutic approaches are mostly based on clinical experience.

The recurrence of FSGS in the transplanted kidney presupposes the presence of one or more circulating factors of extrarenal origin which can selectively affect and damage the glomerular barrier, in particular the podocytes, resulting in massive proteinuria. However, the identity, nature and cellular source of factors circulating in the INS are not yet known.

Recent evidence of the therapeutic efficacy of anti-B cell antibodies in inducing and/or maintaining remission in patients with INS indicates the presence of possible B cell dysfunction.

In support of this, a recent study described the presence of anti-nephrin autoantibodies (a structural component of the podocyte slit diaphragm) in a subgroup of pediatric and adult patients with MCD. These autoantibodies were present during the active phase of the disease, and were associated with a punctate staining of IgG in renal biopsies in correspondence with the specific areas of presence of nephrin. Furthermore, the presence of autoantibodies against nephrin has been found in early post-transplant FSGS recurrence. This preliminary result was confirmed by a Japanese multicenter study conducted on 11 pediatric patients with post-transplant FSGS recurrence. In these patients, anti-nephrin autoantibodies were elevated both before transplantation and during disease relapse and were related to punctate deposition of immunoglobulins G (IgG) that colocalized with nephrin in the graft biopsy at the time of relapse. This recent evidence suggests that circulating anti-nephrin antibodies represent a possible circulating factor involved in the pathogenesis of INS, in particular post-transplant FSGS recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) males and females
* Patients with biopsy-proven idiopathic MCD or FSGS (cases)
* Patients with biopsy-proven idiopathic membranous nephropathy (controls)
* Patients who provided consent to store their samples in the certified CRB biobank

Exclusion Criteria:

* Reasonable possibility of a secondary cause of NS (for cases) or MN (for controls) at time of blood collections
* Active viral or bacterial infections at time of blood collections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the measurement of anti-nephrin antibodies, serum samples stored at the certified Biobank of Rare Diseases and Kidney Diseases of the Mario Negri Pharmacological Research Institute IRCCS from patients with INS (MCD/FSGS) and MN who provided their consent to the conservation of biological samples for future research projects evaluated and authorized by an independent Ethics Committee will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Levels of circulating anti-nephrin autoantibodies | At 1 year. Given the retrospective nature of the study, the indicated time frame refers to the time required to perform the analysis, i.e to assess levels of anti-nephrin antibodies in patients with NS compared to controls.
  Serum samples will be tested for the levels of anti-nephrin autoantibodies by in-house ELISA and results confirmed by commercial ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- Clinical Research Center for Rare Disease Aldo e Cele Daccò, Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCarthy ET, Sharma M, Savin VJ. Circulating permeability factors in idiopathic nephrotic syndrome and focal segmental glomerulosclerosis. Clin J Am Soc Nephrol. 2010 Nov;5(11):2115-21. doi: 10.2215/CJN.03800609. Epub 2010 Oct 21. PMID 20966123
- [Background] D'Agati VD, Kaskel FJ, Falk RJ. Focal segmental glomerulosclerosis. N Engl J Med. 2011 Dec 22;365(25):2398-411. doi: 10.1056/NEJMra1106556. No abstract available. PMID 22187987
- [Background] Gallon L, Leventhal J, Skaro A, Kanwar Y, Alvarado A. Resolution of recurrent focal segmental glomerulosclerosis after retransplantation. N Engl J Med. 2012 Apr 26;366(17):1648-9. doi: 10.1056/NEJMc1202500. No abstract available. PMID 22533598
- [Background] Ruggenenti P, Ruggiero B, Cravedi P, Vivarelli M, Massella L, Marasa M, Chianca A, Rubis N, Ene-Iordache B, Rudnicki M, Pollastro RM, Capasso G, Pisani A, Pennesi M, Emma F, Remuzzi G; Rituximab in Nephrotic Syndrome of Steroid-Dependent or Frequently Relapsing Minimal Change Disease Or Focal Segmental Glomerulosclerosis (NEMO) Study Group. Rituximab in steroid-dependent or frequently relapsing idiopathic nephrotic syndrome. J Am Soc Nephrol. 2014 Apr;25(4):850-63. doi: 10.1681/ASN.2013030251. Epub 2014 Jan 30. PMID 24480824
- [Background] Maas RJ, Deegens JK, Smeets B, Moeller MJ, Wetzels JF. Minimal change disease and idiopathic FSGS: manifestations of the same disease. Nat Rev Nephrol. 2016 Dec;12(12):768-776. doi: 10.1038/nrneph.2016.147. Epub 2016 Oct 17. PMID 27748392
- [Background] Watts AJB, Keller KH, Lerner G, Rosales I, Collins AB, Sekulic M, Waikar SS, Chandraker A, Riella LV, Alexander MP, Troost JP, Chen J, Fermin D, Yee JL, Sampson MG, Beck LH Jr, Henderson JM, Greka A, Rennke HG, Weins A. Discovery of Autoantibodies Targeting Nephrin in Minimal Change Disease Supports a Novel Autoimmune Etiology. J Am Soc Nephrol. 2022 Jan;33(1):238-252. doi: 10.1681/ASN.2021060794. Epub 2021 Nov 3. PMID 34732507
- [Background] Casiraghi F, Todeschini M, Podesta MA, Mister M, Ruggiero B, Trillini M, Carrara C, Diadei O, Villa A, Benigni A, Remuzzi G. Immunophenotypic Alterations in Adult Patients with Steroid-Dependent and Frequently Relapsing Nephrotic Syndrome. Int J Mol Sci. 2023 Apr 22;24(9):7687. doi: 10.3390/ijms24097687. PMID 37175393
- [Background] Salfi G, Casiraghi F, Remuzzi G. Current understanding of the molecular mechanisms of circulating permeability factor in focal segmental glomerulosclerosis. Front Immunol. 2023 Sep 19;14:1247606. doi: 10.3389/fimmu.2023.1247606. eCollection 2023. PMID 37795085
- [Background] Shirai Y, Miura K, Ishizuka K, Ando T, Kanda S, Hashimoto J, Hamasaki Y, Hotta K, Ito N, Honda K, Tanabe K, Takano T, Hattori M. A multi-institutional study found a possible role of anti-nephrin antibodies in post-transplant focal segmental glomerulosclerosis recurrence. Kidney Int. 2024 Mar;105(3):608-617. doi: 10.1016/j.kint.2023.11.022. Epub 2023 Dec 16. PMID 38110152